CLINICAL TRIAL: NCT03517280
Title: The Role of Nutritional Status in the Treatment of Neuroblastoma
Brief Title: Nutritional Status in Neuroblastoma in Sao Paolo, Brazil
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Instituto de Tratamento do Câncer Infantil (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR7865
Record Dates: First submitted 2018-03-14; First posted 2018-05-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Neuroblastoma
Keywords: Malnutrition; Childhood Cancer; Nutrition Aspect of Cancer; Child Malnutrition; Brazil; Sao Paolo
MeSH Terms: conditions — Neuroblastoma; Malnutrition; Neoplasms; Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection to bank plasma and serum will occur at diagnosis, after completion of immune therapy and at 12 month post-treatment.
  For micronutrient analysis, 3 to 5 mL of the patient's venous blood will be collected without anticoagulant to study To obtain serum and plasma, to bank for future micronutrient analysis, blood samples (10 mL) will be collected by venipuncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Neuroblastoma: Children undergoing treatment for Neuroblastoma at ITACI in Sao Paolo in Brazil who are under the age of 18 years.

SUMMARY:
This study proposes to investigate the effect of treatment of neuroblastoma on nutritional status, assessed by body mass index (BMI) z score, and body composition evaluated by mid-upper arm circumference (MUAC), from diagnosis through 1-year post end of treatment. The study also aims to investigate the nutritional status and its role in toxicities, infection, survival rates, disease relapse, cost of care and readmission rates, as well as health-related quality of life. The study will take place in Sao Paolo in Brazil, where an estimated sample of 50 children with neuroblastoma will be recruited for the period of 2 years.

DETAILED DESCRIPTION:
In Brazil, cancer represents the leading cause of death by disease in children and adolescents from 1 to 19 years old. Neuroblastomas correspond to nearly 10% of all cancer diagnoses among children younger than 15 years of age, with an incidence of 1 case per 100,000 children of this age group. About 500 new cases of neuroblastoma (NB) are diagnosed annually in Brazil. The complexity and intensity of treatment result in several treatment-related toxicities (TRT) that make it challenging to maintain nutritional status in these nutritionally at-risk patients. In Brazil, up to 26% of undernutrition at diagnosis has been found in patients with solid tumors. In neuroblastoma, high prevalence rates of malnutrition have been reported elsewhere with up to 80% of children at diagnosis and 20-50% during treatment classified as undernourished. It's important to underscore that nutritional status is a modifiable risk factor, therefore it needs more attention and close monitoring. It is important to better comprehend the effect of treatment for neuroblastoma on nutritional status and body composition, for which prospective longitudinal studies are required. Therefore, in this prospective cohort study, the investigators will evaluate the fluctuations in nutritional status over the course of treatment in children with neuroblastoma at the study center in São Paulo, Brazil. The results of this study will drive the development of evidence-based guidelines for the nutritional care of children with neuroblastoma and set research priorities for subsequent investigations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high-risk neuroblastoma at ITACI, according to the Pediatric Oncology Group (POG)/Children's Cancer Study Group (CCG) classification (International Neuroblastoma Staging System (INSS) stage)
* Age under 18 years
* Informed consent from a legal guardian to participate in the study

Exclusion Criteria:

* Patients who have received previous chemotherapy
* First assessment performed more than 48 hours after the beginning of treatment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Demographic variables will be collected from medical records, including date of birth, sex, city/state/country of residence, date of diagnosis and ethnicity. Socioeconomic data (per capita annual income and living conditions) will be drawn from the institutions' social work service charts. The data will be collected in hospital - Instituto de Tratamento do Câncer Infantil, in Sao Paolo, Brazil.
  The investigators will also collect clinical outcome data from the medical chart. The incidence of infectious toxicity, all Grade 3 and 4 toxicities (defined by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC)), death, disease relapse or progression, number of days in the hospital and delays in treatment will be documented during each cycle.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Body Mass Index Z Score | Up to 1 year post treatment
  Effect of neuroblastoma treatment in nutritional status: Nutritional status will be measured by BMI Z score
Mid-upper arm circumference (MUAC) | Up to 1 year post treatment
  Effect of neuroblastoma treatment in body composition: Body composition will be measured by mid-upper arm circumference (MUAC)
Measurement from Bioelectrical Impedance Analysis (BIA) | Up to 1 year post treatment
  Effect of neuroblastoma treatment in body composition: Body composition will be measured by BIA

SECONDARY OUTCOMES:
Cumulative number of Grade 3/4 toxicities | 2 years
  Investigate association of nutritional status and the occurrence of grade 3/4 toxicities using NCI Common Toxicity Criteria (CTC)
Incidence of newly diagnosed infection | 2 years
  Study the association of nutritional status and infection classified from moderate to severe neutropenia (ANC < 500)
Survival rate | Up to 1 year post treatment
  Survival is defined by both overall survival (time from enrollment to death from any cause) and event-free survival (time from enrollment to the first episode of relapse, disease progression or death).
Disease relapse rate | Up to 1 year post treatment
  Investigate the association of nutritional status and disease relapse
Cost of care | Up to 1 year post treatment
  Investigate the association of nutritional status and the cost of care defined by the sum of the cost of duration of hospital stay and cost of readmission rates. We will evaluate the values individually and collectively.
Score on HuPS or HUI | Up to 1 year post treatment
  Health-related quality of life will be measured by the Health Utilities Preschool(HuPS) survey for 2 -5 years old or by Health Utilities Index (HUI) for 5 years and older (assessment is not considered for children under 2 years), during and after treatment, and its association with nutritional status and body composition. These are complementary instruments for use in the contiguous age groups. They are scored in the same way.
Score on 24-hour Dietary Recalls | Up to 1 year post treatment
  Investigate the association of nutritional status and diet quality, measured by 24h dietary recalls

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ladas, Phd, RD, Study Director — Columbia University; Karina Viani, RD, Principal Investigator — Instituto de Tratamento do Câncer Infantil, Sao Paolo; Vicente Odone, MD, PhD, Study Chair — Instituto de Tratamento do Câncer Infantil, Sao Paolo
Locations (1):
- Instituto de Tratamento do Câncer Infantil, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The database is secured in Brazil research site at ITACI. De-identified data is shared with Columbia University Medical Center via REDCap database system - managed by Columbia University